CLINICAL TRIAL: NCT05850624
Title: Effect of Virtual Reality Animation and Ice Massage on The Hoku Point on Labor Pain, Duration of Labor, and Satisfaction
Brief Title: Virtual Reality Animation and Ice Massage on The Hoku Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Şahika ŞİMŞEK ÇETİNKAYA, Head of Midwifery, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-KAEK-53
Record Dates: First submitted 2023-04-03; First posted 2023-05-09 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Labor Pain
Keywords: birth pain,; satisfaction; ice massage; virtual reality
MeSH Terms: conditions — Labor Pain; Personal Satisfaction | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ice massage (Experimental): ice massage to hoku point for labor pain for 20 minutes
  Interventions: Other: ice massage
- virtual animation (Experimental): watching virtual animation for 20 minutes for labor pain
  Interventions: Other: virtual reality animation
- Control Group (No Intervention): receiving standart care

INTERVENTIONS:
Other: ice massage — active phase when cervical dilatation was 6-8 cm. Ice will apply to the huko point (LI4 area) which is located on the dorsum of the hand, between the first and second metacarpal bones, between the thumb and the index finger for 20 minutes with an ice pack
  Other Names: supportive care
  Arms: ice massage
Other: virtual reality animation — cervical dilatation was 6-8 cm. Immediately after the second VAS application, the women will be asked about the video they wanted to watch of the sound of waves in the Ocean, rain falling or blooming trees with virtual reality glass. animation will show for a total of 20 min.
  Other Names: supportive care
  Arms: virtual animation

SUMMARY:
The goal of this study was to compare the effects of ice massage and virtual reality animation on labor pain, duration, and satisfaction with delivery.

The main questions aims to answer are:

H1 There are differences between Ice massage group and/or virtual reality animation groups and the control group in women's' labor pain.

H2 There are differences between Ice massage group and/or virtual reality animation groups and the control group in women's' labor duration.

H3 There are differences between Ice massage group and/or virtual reality animation groups and the control group in women's' satisfaction.

This randomized controlled trial (n = 94) includes three arms. Two intervention groups (ice massage (IMG); virtual reality animation (VRA)) and one control group, (CG). Personal information form, and Visual Analog Scale (VAS) and Birth Satisfaction Scale will used to collect data. Frequency and percentage calculations, Mann Whitney U, Kruskal Wallis test, chi-square test, Tukey's honestly significant difference test, and will used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Term primiparous and singleton pregnancies,
* Longitudinal and vertex position of the fetus,
* Body Mass Index (BMI) below 30,
* cervical dilatation of 0-3 cm,
* who agreed to participate in the study

Exclusion Criteria:

* applying pharmacological intervention during labor,
* having a risky pregnancy,
* want to withdraw from the study,
* having ice allergy,
* being visually impaired.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
labor pain | "Change from Baseline cervical dilatation 0-3 cm (duration can change 8-9 hours)
  Visual Analogue Scale (VAS)I
labor duration | "Change from Baseline cervical dilatation 6-8 cm(duration can change 4-8 hours)
  Personal Information Form
labor duration | hour of latent phase ( duration can change 8-9 hour)
  Personal Information Form
labor duration | hour of placental expulsion (duration can change 10 minutes to 30 minutes)
  Personal Information Form
birth satisfaction | postpartum period up to 24 hours
  Birth Satisfaction Scale - Revised (BSS-R)
labor pain | active phase up to 20 hours
  Visual Analogue Scale (VAS) II
labor duration | hour of total delivery (can change 14-18 hours)
  Personal Information Form

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I do not want to make individual participant data (IPD) available to other researchers.